CLINICAL TRIAL: NCT06052995
Title: Observational Study to Evaluate the Actual Use of Elidel® in South and East Asian Patients From 3 Months to 12 Years With Mild to Moderate Atopic Dermatitis.
Brief Title: Observational Study to Evaluate Use of Elidel® in South and East Asian Pediatric Patients With Atopic Dermatitis.
Acronym: Elidel-SEA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MEDA PHARMA SPA, a Viatris company (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: PCLS-CRZ-4001
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Mild to Moderate Atopic Dermatitis
MeSH Terms: interventions — pimecrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Elidel 1% Topical Cream — Elidel® 1% is a non-steroid cream for cutaneous use containing pimecrolimus. It is indicated for mild or moderate AD.

SUMMARY:
Elidel® is indicated for the short-term treatment and long-term management of signs and symptoms of atopic dermatitis (AD) in infants (3 to 23 months), children (2 to 11 years), adolescents (12 to 17 years), and adults. However, little evidence is available in literature in South and East Asian population. Hence, this non interventional study (NIS) is designed to capture data about the actual use of Elidel® in South and East Asian patients from 3 months to 12 years with mild to moderate AD.

DETAILED DESCRIPTION:
Once the clinical decision has been made to prescribe Elidel® to a patient according to the local Package Insert, the investigator will consider recruiting the patient into this NIS. The decision to prescribe Elidel® must be prior to and independent from the decision to include the patient into the NIS.

As per study design:

* Visit 1 (V1; Inclusion): Only after the decision of prescribing Elidel® has been made, eligible patients will be asked for their agreement to participate in the study.
* V1a/b/c (optional visits): AD related visits between Inclusion and Elidel® Treatment Interruption - according to routine clinical practice
* Visit 2 (V2; Elidel® Treatment Interruption): Investigators will decide to interrupt Elidel® treatment because of success or failure: Treatment success: Patient's symptoms improved and does not need to continue the Elidel® treatment. Treatment failure: Patient's symptoms worsened and need to switch to a different treatment.
* V2a/b/c (optional visits): AD related follow-up visits between Elidel® Treatment Interruption and EOS - According to routine clinical practice.
* Visit 3 (V3; End of Study): The study ends after the Maintenance Period of at least 3 months allowing certain flexibility to respond to the routine practice.

End of Study will be approximately 6 months after the inclusion depending on length of the Elidel® Treatment Period. Collection of data includes but not limited to patients' demographics, clinical history, clinical symptom and manifestation, comorbidities, reported adverse events and concomitant medications. The patients' questionnaires (IDQOL and CDLQI) will be utilized to collect data directly from enrolled patients and transferred into the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility should be reviewed and documented by an appropriately qualified member of the investigator's study team before patients are included in the study.

Patients must meet all of the following inclusion criteria to be eligible for enrolment into the study:

* Patients that have been prescribed Elidel® according to the local Package Insert prior to and independently from patient's enrolment into the study.
* Patients of Asian ethnicity
* Patients within following age group for respective countries as defined below:

Malaysia: Patients > 2 years and <12 years old. Hong Kong: Patients >3 months and <12 years old. Thailand: Patients >3 months and <12 years old. Taiwan: Patients >3 months and <12 years old.

* Signed informed consent from patient and (as per local regulations) if applicable from parent(s) or legal guardian(s) in compliance with local requirements
* Patients with mild to moderate AD (SCORAD Index <50)

Exclusion Criteria:

Patient candidates must not be enrolled in the study if they meet any of the following criteria:

* Patients for whom Elidel® is not recommended accordingly to the local Package Insert
* Patients with severe AD (SCORAD Index ≥50)
* Receiving systemic glucocorticoids, antibiotics, antifungals, immunomodulators, antihistamines and ultraviolet radiation therapy within the last 4 weeks before inclusion
* Receiving any topical AD-effective drugs within the last 2 weeks before inclusion
* Pregnant and/or breastfeeding women
* Patients or parent(s) / legal guardian (as applicable) that are not able to fulfil study requirements according to investigator's opinion
* Patients or parent(s) / legal guardian (as applicable) that refuse to participate to the study

Ages: 3 Months to 12 Years | Sex: All
Age Groups: Child
Study Population: Approximately 130 patients will be enrolled.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
SCORAD Change | 6 months
  SCORing Atopic Dermatitis (SCORAD) Index change in the Atopic Dermatitis (AD) areas from inclusion to the end of Elidel® treatment period (V2)

SECONDARY OUTCOMES:
Treatment Duration | 6 months
  Treatment duration with Elidel®
Reduction of symptoms over time | 6 months
  Reduction of symptoms (itching and sleep loss) during Elidel® treatment period based on the Visual Analogue Scale (VAS) in the SCORAD index.
Number of days lost | 6 months
  Number of days lost from school and/or work for patients and/or caregivers, assessed at each visit.
Adverse events over time | 6 months
  Elidel® safety and tolerability (adverse drug reactions [ADRs] and special situations [SpS]) during the whole study period.